CLINICAL TRIAL: NCT05621304
Title: Optimizing HBV Care Cascade Among Foreign-Born in the United States (FOCUS-HBV Study)
Status: Recruiting | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10001125; 001125-DK
Record Dates: First submitted 2022-11-16; First posted 2022-11-18 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-05-14

CONDITIONS: Chronic Hepatitis B Virus (Hbv)
Keywords: Healthcare Retention; Natural History; Acculturation-Related Barriers
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Foreign Born subjects w/Chronic HBV: foreign born (FB) chronic hepatitis B subjects

SUMMARY:
Background:

People who were born outside of the country are the largest group of adults infected with chronic hepatitis B virus (HBV) in the US. HBV affects the liver. If not treated, HBV infection can lead to serious liver disease, including cancer. One recent study showed that only 35% of foreign-born US adults were aware of their HBV infections. Foreign-born US adults may also have trouble getting proper care after they are diagnosed with HBV. In one small survey, language, cultural, and financial barriers were cited as the biggest reasons for not receiving care. To help more people with HBV, researchers want to learn how to find and overcome any barriers to care.

Objective:

This natural history study seeks to identify and better understand barriers that prevent foreign-born US adults from getting proper care for HBV infections.

Eligibility:

People aged 18 years and older with chronic HBV who were born outside of the US.

Design:

Participants will visit the NIH clinic 1 time. This visit will take about 20 minutes.

Researchers will review participants medical records and collect information about their HBV.

Participants will complete a survey. They will answer questions about:

Where they came from.

When they came to the US.

How well they have adapted to living in the US.

The health care they have received for HBV.

Their age, gender, and education.

Participants will be paid $10 for completing the survey.

DETAILED DESCRIPTION:
Study Description:

This is an observational, prospective study in which Foreign-Born (FB) participants with chronic hepatitis B virus (HBV) will be consented and then surveyed to better understand and identify acculturation-related barriers in the HBV care cascade and to optimize healthcare retention for those with HBV.

Objectives:

Primary Objective:

-To assess the association between recent immigration (defined by less than 10 years length of residence in US) and progression through the HBV care cascade post-diagnosis among foreign-born diagnosed with chronic HBV infection.

Secondary Objectives:

* To characterize and quantify completion of HBV care metrics after diagnosis (both proportion and time to completion) for a multi-ethnic cohort of foreign-born adults
* To compare gaps in completion of post-diagnosis care metrics by recent immigrant status and racial/ethnic group
* To develop and pilot a multi-national survey instrument to accurately and reliably measure immigration-related factors
* To determine impact of immigration-related factors (e.g. acculturation, language proficiency, region of origin) on completion of care metrics overall and among recent immigrants

Endpoints:

Primary Endpoint:

-The primary endpoint is to assess the proportion of FB diagnosed with HBV who have completed an initial visit for diagnosis of chronic HBV infection (defined as a visit with either primary or specialty provider during which testing for treatment eligibility was ordered).

Secondary Endpoints:

* Completion of testing to determine eligibility for treatment

  * Minimum sufficient set of labs including hepatitis B e-antigen (HBeAg), ALT, HBV DNA, and HIV testing
  * Fibrosis assessment which can be non-invasive (FIB-4/APRI, US elastography or MR elastography) or invasive (liver biopsy)
* Treatment uptake if eligible based on AASLD guidelines on treatment eligibility

  * HBV DNA>2000 IU/mL and ALT>2x ULN if HBeAgnegative
  * HBV DNA>20000 IU/mL and ALT>2x ULN if HBeAgpositive
  * Cirrhosis or HCC
  * Family history of HCC
* Retention in care

  * At least annual visit for HBV diagnosis with appropriate lab tests ordered
  * Ultrasound and AFP for HCC surveillance screening for those who are indicated

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Male or female, aged >=18 years
* Diagnosed of chronic HBV (HBsAg-positive)
* Self-reported country of birth outside of the US

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

-Individuals not able to understand and sign the informed consent document will not be included in the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Foreign Born subjects with Chronic HBV
Sampling Method: Non-Probability Sample
Enrollment: 255 (Estimated)
Dates: Start 2017-01-03 (Actual); Primary Completion 2026-12-29 (Estimated); Study Completion 2026-12-29 (Estimated)

PRIMARY OUTCOMES:
Assess the association between recent immigration (defined by less than 10 years length of residence in US) and progression through the HBV care cascade post-diagnosis among foreign-born diagnosed with chronic HBV infection | Visit 1
  The reason for this distinction is to separate visits for screening from linkage to care, which may in some clinics occur with the same provider.

CONTACTS AND LOCATIONS:
Overall Officials: Christine C Hsu, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (2):
- United States (2):
  - University of Southern California, Los Angeles, California
  - National Institutes of Health Clinical Center, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001125-DK.html